CLINICAL TRIAL: NCT03426358
Title: Usefulness of Liver Stiffness Measurement in Predicting Hepatic Veno-Occlusive Disease Development in Patients Who Undergo HSCT: a Multicentric Prospective Study
Brief Title: Liver Stiffness Measurement Predicts VOD/SOS Development (ELASTOVOD ITALIAN MULTICENTRIC STUDY)
Acronym: ELASTOVOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Davide Festi, Principal Investigator (PI), IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ELASTOVOD
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Veno Occlusive Disease, Hepatic; Sinusoidal Obstruction Syndrome; Stem Cell Transplant Complications
Keywords: Veno Occlusive Disease; Sinusoidal Obstruction Syndrome; HSCT; Hematopoietic Stem Cell Transplantation; Stem Cell Transplant Complications; Liver Stiffness Measurement; Sinusoidal Obstructive Syndrome; Transient Elastography
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Intervention Model Description: All the patients with onco-hematological disease and an indication for transplantation of hematopoietic stem cells will be consecutively studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing HSCT (Experimental): LSM assessed by Elastographic Techniques
  Interventions: Device: LSM assessed by Elastographic Techniques

INTERVENTIONS:
Device: LSM assessed by Elastographic Techniques — Performing Transient Elastography, ARFI or 2D-SWE on patients at baseline (within 1 month before HSCT) and after HSCT on days +9/10, +15/17, +22/24

SUMMARY:
ELASTOVOD is a prospective multicenter study, involving several centers of Onco-haematology in Italy. Investigators perform hepatic elastographic measurements (with Transient Elastography, ARFI or 2D-SWE) on patients undergoing HSCT, at baseline before transplantation (T0) and at T1/T2/T3 after HSCT (+9/10, +15/17, +22/24).

SOS/VOD diagnosis was performed according to clinical criteria.

DETAILED DESCRIPTION:
Sinusoidal Obstruction Syndrome (SOS), also known as hepatic Veno-Occlusive Disease (VOD), is a life-threatening complication in patients undergoing Hematopoietic Stem Cells Transplantation (HSCT) for onco-haematological disease.

In the severe form, mortality rate can be high as 80%. Patients developing SOS/VOD present a higher survival rate when earlier SOS/VOD- specific therapy has initiated. In order to get better outcomes, it is necessary to improve early diagnosis of SOS/VOD, finding new non--invasive diagnostic instruments.

The aim of this prospective multicenter study is to assess in a large, mixed (adult and paediatric) population undergoing HSCT, the diagnostic role for SOS/VOS of Liver Stiffness Measurement (LSM), assessed by different elastographic methods.

In our study, Liver Stiffness Measurement (LSM) can be measured by Transient Elastography (TE) with Fibroscan, Acoustic Radiation Force Impulse (ARFI) or 2D-Share Wave Elastography (2D-SWE). Once chosen an elastometric method at baseline, the same must be used for all subsequent evaluations of the patient.

In patients undergoing HSCT, within one month, a complete baseline evaluation is provided. Baseline evaluation (T0) includes: signature of informed consent, haematological and hepatological anamnesis, in order to assess comorbidities and risk factors for hepato-biliary complications; complete laboratory tests; abdominal Color-Doppler Ultrasound and hepatic Elastography (with Transient Elastography, ARFI or 2D-SWE).

After conditioning and HSCT, each patient is evaluated at T1 (+9/10), T2 (+15/17), T3 (+22/24) with: bedside Elastography, laboratory tests, clinical examination based on clinical criteria for SOS/VOD diagnosis (e.g. Baltimora criteria, modified Seattle criteria, new EBMT criteria).

RUCAM-CIOMS Scale can be assess, in order to establish DILI (Drug Induced Liver Injury) diagnosis, as well.

In case of SOS/VOD suspicion, patient goes through an intense monitoring period: laboratory tests, clinical evaluation for SOS/VOD diagnosis, Color-Doppler US and Elastography are repeatedly performed in next days. This monitoring period stops if diagnosis of SOS/VOD or other diagnosis is reached.

Each center will prospectively collect data according to an electronic e-CFR on REDCap (Research Electronic Data Capture) system, a web application designed to support data capture for research studies in a secure manner.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* age between 3 and 70
* patients suffering from an onco-hematological disease that have an indication for either allogenic or autologous hematopoietic stem cells transplantation
* obtaining of informed consent

Exclusion Criteria:

* pathological obesity (BMI >40)
* pacemaker of implantable defibrillator
* presence of ascites at baseline

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic Role of Liver Stiffness Measurement in SOS/VOD development | From HSCT to 30 days after HSCT
  To assess in a large, mixed (adult and paediatric) population undergoing HSCT, the role of Liver Stiffness Measurement (LSM), assessed by different elastographic methods, in SOS/VOD diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colecchia, M.D., Principal Investigator — Azienda Ospedaliera-Universitaria Integrata di Verona; Francesca Bonifazi, Ph.D. M.D., Study Chair — Azienda Ospedaliera-Universitaria Sant'Orsola Malpighi di Bologna; Andrea Passion, Prof. M.D., Study Chair — Azienda Ospedaliera-Universitaria Sant'Orsola Malpighi di Bologna
Locations (37):
- Italy (37):
  - Azienda Ospedaliera Universitaria di Bologna Policlinico S. Orsola Malpighi., Bologna, BO
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera "Card. G. Panico", Tricase, Lecce
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Policlinico Umberto I - Università la Sapienza, Roma, RM
  - Azienda Ospedaliera-Nazionale SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero-Universitaria Consorziale - Policlinico di Bari, Bari
  - ASST Papa Giovanni XXIII Ospedali riuniti di Bergamo, Bergamo
  - Azienda Sanitaria dell'Alto Adige, Bolzano
  - Spedali Civili di Brescia, UO Ematologia, Brescia
  - Policlinico Vittorio Emanuele - Presidio Ferrarotto, Catania
  - Azienda Ospedaliera-Universitaria Careggi, Florence
  - Azienda Ospedaliera-Universitaria Meyer, Florence
  - Ospedale Policlinico San Martino, Genova
  - Ospedale Vito Fazzi, Lecce
  - Ospedale dell'Angelo, Mestre
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Maggiore Policlinico di Milano, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera-Universitaria di Modena, Modena
  - Ospedale Pediatrico Pausilipon, Napoli
  - Policlinico Federico II, Napoli
  - Azienda Ospedaliero-Universitaria di Padova, Padua
  - Azienda Ospedaliera Ospedali riuniti Villa Sofia- Cervello, Palermo
  - Azienda Ospedaliero-Universitaria Ospedale Maggiore di Parma, Parma
  - Azienda Sanitaria Locale di Pescara, Pescara
  - Azienda Ospedaliero-universitaria Pisana, UO Ematologia, Pisa
  - Azienda Ospedaliero-Universitaria Pisana, UO Oncoematologia Pediatrica, Pisa
  - Arcispedale S. Maria Nuova di Reggio Emilia, Reggio Emilia
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Policlinico Tor Vergata, Roma
  - Policlinico Universitario A. Gemelli, Roma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza, Torino
  - Azienda Ospedaliero-Universitaria Integrata di Udine, Udine
  - Azienda Ospedaliero-Universitaria Integrata di Verona, Verona
  - Azienda Ospedaliera di Vicenza, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wadleigh M, Ho V, Momtaz P, Richardson P. Hepatic veno-occlusive disease: pathogenesis, diagnosis and treatment. Curr Opin Hematol. 2003 Nov;10(6):451-62. doi: 10.1097/00062752-200311000-00010. PMID 14564177
- [Background] McDonald GB. Hepatobiliary complications of hematopoietic cell transplantation, 40 years on. Hepatology. 2010 Apr;51(4):1450-60. doi: 10.1002/hep.23533. PMID 20373370
- [Background] Carreras E, Diaz-Beya M, Rosinol L, Martinez C, Fernandez-Aviles F, Rovira M. The incidence of veno-occlusive disease following allogeneic hematopoietic stem cell transplantation has diminished and the outcome improved over the last decade. Biol Blood Marrow Transplant. 2011 Nov;17(11):1713-20. doi: 10.1016/j.bbmt.2011.06.006. Epub 2011 Jun 25. PMID 21708110
- [Background] Jones RJ, Lee KS, Beschorner WE, Vogel VG, Grochow LB, Braine HG, Vogelsang GB, Sensenbrenner LL, Santos GW, Saral R. Venoocclusive disease of the liver following bone marrow transplantation. Transplantation. 1987 Dec;44(6):778-83. doi: 10.1097/00007890-198712000-00011. PMID 3321587
- [Background] McDonald GB, Sharma P, Matthews DE, Shulman HM, Thomas ED. Venocclusive disease of the liver after bone marrow transplantation: diagnosis, incidence, and predisposing factors. Hepatology. 1984 Jan-Feb;4(1):116-22. doi: 10.1002/hep.1840040121. PMID 6363247
- [Background] Mohty M, Malard F, Abecassis M, Aerts E, Alaskar AS, Aljurf M, Arat M, Bader P, Baron F, Bazarbachi A, Blaise D, Ciceri F, Corbacioglu S, Dalle JH, Dignan F, Fukuda T, Huynh A, Masszi T, Michallet M, Nagler A, NiChonghaile M, Okamoto S, Pagliuca A, Peters C, Petersen FB, Richardson PG, Ruutu T, Savani BN, Wallhult E, Yakoub-Agha I, Duarte RF, Carreras E. Revised diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in adult patients: a new classification from the European Society for Blood and Marrow Transplantation. Bone Marrow Transplant. 2016 Jul;51(7):906-12. doi: 10.1038/bmt.2016.130. Epub 2016 May 16. PMID 27183098
- [Background] Corbacioglu S, Carreras E, Ansari M, Balduzzi A, Cesaro S, Dalle JH, Dignan F, Gibson B, Guengoer T, Gruhn B, Lankester A, Locatelli F, Pagliuca A, Peters C, Richardson PG, Schulz AS, Sedlacek P, Stein J, Sykora KW, Toporski J, Trigoso E, Vetteranta K, Wachowiak J, Wallhult E, Wynn R, Yaniv I, Yesilipek A, Mohty M, Bader P. Diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in pediatric patients: a new classification from the European society for blood and marrow transplantation. Bone Marrow Transplant. 2018 Feb;53(2):138-145. doi: 10.1038/bmt.2017.161. Epub 2017 Jul 31. PMID 28759025
- [Background] Dignan FL, Wynn RF, Hadzic N, Karani J, Quaglia A, Pagliuca A, Veys P, Potter MN; Haemato-oncology Task Force of British Committee for Standards in Haematology; British Society for Blood and Marrow Transplantation. BCSH/BSBMT guideline: diagnosis and management of veno-occlusive disease (sinusoidal obstruction syndrome) following haematopoietic stem cell transplantation. Br J Haematol. 2013 Nov;163(4):444-57. doi: 10.1111/bjh.12558. Epub 2013 Sep 17. PMID 24102514
- [Background] Sorror ML, Maris MB, Storb R, Baron F, Sandmaier BM, Maloney DG, Storer B. Hematopoietic cell transplantation (HCT)-specific comorbidity index: a new tool for risk assessment before allogeneic HCT. Blood. 2005 Oct 15;106(8):2912-9. doi: 10.1182/blood-2005-05-2004. Epub 2005 Jun 30. PMID 15994282
- [Background] Richardson PG, Smith AR, Triplett BM, Kernan NA, Grupp SA, Antin JH, Lehmann L, Miloslavsky M, Hume R, Hannah AL, Nejadnik B, Soiffer RJ. Earlier defibrotide initiation post-diagnosis of veno-occlusive disease/sinusoidal obstruction syndrome improves Day +100 survival following haematopoietic stem cell transplantation. Br J Haematol. 2017 Jul;178(1):112-118. doi: 10.1111/bjh.14727. Epub 2017 Apr 26. PMID 28444784
- [Background] Berzigotti A, Castera L. Update on ultrasound imaging of liver fibrosis. J Hepatol. 2013 Jul;59(1):180-2. doi: 10.1016/j.jhep.2012.12.028. Epub 2013 Jan 15. No abstract available. PMID 23333447
- [Background] Lassau N, Auperin A, Leclere J, Bennaceur A, Valteau-Couanet D, Hartmann O. Prognostic value of doppler-ultrasonography in hepatic veno-occlusive disease. Transplantation. 2002 Jul 15;74(1):60-6. doi: 10.1097/00007890-200207150-00011. PMID 12134100
- [Background] Lassau N, Leclere J, Auperin A, Bourhis JH, Hartmann O, Valteau-Couanet D, Benhamou E, Bosq J, Ibrahim A, Girinski T, Pico JL, Roche A. Hepatic veno-occlusive disease after myeloablative treatment and bone marrow transplantation: value of gray-scale and Doppler US in 100 patients. Radiology. 1997 Aug;204(2):545-52. doi: 10.1148/radiology.204.2.9240551.
- [Background] Karlas T, Weber J, Nehring C, Kronenberger R, Tenckhoff H, Mossner J, Niederwieser D, Troltzsch M, Lange T, Keim V. Value of liver elastography and abdominal ultrasound for detection of complications of allogeneic hemopoietic SCT. Bone Marrow Transplant. 2014 Jun;49(6):806-11. doi: 10.1038/bmt.2014.61. Epub 2014 Apr 7. PMID 24710567
- [Background] Auberger J, Graziadei I, Clausen J, Vogel W, Nachbaur D. Non-invasive transient elastography for the prediction of liver toxicity following hematopoietic SCT. Bone Marrow Transplant. 2013 Jan;48(1):159-60. doi: 10.1038/bmt.2012.113. Epub 2012 Jun 18. No abstract available. PMID 22705804
- [Background] Sandrin L, Fourquet B, Hasquenoph JM, Yon S, Fournier C, Mal F, Christidis C, Ziol M, Poulet B, Kazemi F, Beaugrand M, Palau R. Transient elastography: a new noninvasive method for assessment of hepatic fibrosis. Ultrasound Med Biol. 2003 Dec;29(12):1705-13. doi: 10.1016/j.ultrasmedbio.2003.07.001. PMID 14698338
- [Background] Fontanilla T, Hernando CG, Claros JC, Bautista G, Minaya J, Del Carmen Vega M, Piazza A, Mendez S, Rodriguez C, Aranguena RP. Acoustic radiation force impulse elastography and contrast-enhanced sonography of sinusoidal obstructive syndrome (Veno-occlusive Disease): preliminary results. J Ultrasound Med. 2011 Nov;30(11):1593-8. doi: 10.7863/jum.2011.30.11.1593. PMID 22039033
- [Background] Bureau C, Metivier S, Peron JM, Selves J, Robic MA, Gourraud PA, Rouquet O, Dupuis E, Alric L, Vinel JP. Transient elastography accurately predicts presence of significant portal hypertension in patients with chronic liver disease. Aliment Pharmacol Ther. 2008 Jun;27(12):1261-8. doi: 10.1111/j.1365-2036.2008.03701.x. Epub 2008 Apr 4. PMID 18397389
- [Background] Bota S, Herkner H, Sporea I, Salzl P, Sirli R, Neghina AM, Peck-Radosavljevic M. Meta-analysis: ARFI elastography versus transient elastography for the evaluation of liver fibrosis. Liver Int. 2013 Sep;33(8):1138-47. doi: 10.1111/liv.12240. Epub 2013 Jul 16. PMID 23859217
- [Background] Millonig G, Reimann FM, Friedrich S, Fonouni H, Mehrabi A, Buchler MW, Seitz HK, Mueller S. Extrahepatic cholestasis increases liver stiffness (FibroScan) irrespective of fibrosis. Hepatology. 2008 Nov;48(5):1718-23. doi: 10.1002/hep.22577. PMID 18836992
- [Background] Bamber J, Cosgrove D, Dietrich CF, Fromageau J, Bojunga J, Calliada F, Cantisani V, Correas JM, D'Onofrio M, Drakonaki EE, Fink M, Friedrich-Rust M, Gilja OH, Havre RF, Jenssen C, Klauser AS, Ohlinger R, Saftoiu A, Schaefer F, Sporea I, Piscaglia F. EFSUMB guidelines and recommendations on the clinical use of ultrasound elastography. Part 1: Basic principles and technology. Ultraschall Med. 2013 Apr;34(2):169-84. doi: 10.1055/s-0033-1335205. Epub 2013 Apr 4. PMID 23558397
- [Background] Lucena MI, Garcia-Cortes M, Cueto R, Lopez-Duran J, Andrade RJ. Assessment of drug-induced liver injury in clinical practice. Fundam Clin Pharmacol. 2008 Apr;22(2):141-58. doi: 10.1111/j.1472-8206.2008.00566.x. Erratum In: Fundam Clin Pharmacol. 2009 Feb;23(1):147. PMID 18353109
- [Background] del Campo L, Leon NG, Palacios DC, Lagana C, Tagarro D. Abdominal complications following hematopoietic stem cell transplantation. Radiographics. 2014 Mar-Apr;34(2):396-412. doi: 10.1148/rg.342135046. PMID 24617687
- [Background] Mohty M, Malard F, Abecassis M, Aerts E, Alaskar AS, Aljurf M, Arat M, Bader P, Baron F, Bazarbachi A, Blaise D, Ciceri F, Corbacioglu S, Dalle JH, Duarte RF, Fukuda T, Huynh A, Masszi T, Michallet M, Nagler A, NiChonghaile M, Pagluica T, Peters C, Petersen FB, Richardson PG, Ruutu T, Savani BN, Wallhult E, Yakoub-Agha I, Carreras E. Sinusoidal obstruction syndrome/veno-occlusive disease: current situation and perspectives-a position statement from the European Society for Blood and Marrow Transplantation (EBMT). Bone Marrow Transplant. 2015 Jun;50(6):781-9. doi: 10.1038/bmt.2015.52. Epub 2015 Mar 23. PMID 25798682
- [Background] Colecchia A, Marasco G, Ravaioli F, Kleinschmidt K, Masetti R, Prete A, Pession A, Festi D. Usefulness of liver stiffness measurement in predicting hepatic veno-occlusive disease development in patients who undergo HSCT. Bone Marrow Transplant. 2017 Mar;52(3):494-497. doi: 10.1038/bmt.2016.320. Epub 2016 Dec 12. No abstract available. PMID 27941774
- [Derived] Ravaioli F, Colecchia A, Peccatori J, Pagliara D, Grassi A, Barbato F, Masetti R, Sarina B, Sica S, Cesaro S, Nozzoli C, Assanto GM, Prezioso L, Santarone S, Saglio F, Vanni E, Olivieri A, Delia M, Benedetti E, Zallio F, Pane F, Skert C, Menconi M, Benedetti F, De Felice F, Colecchia L, Belotti T, Alemanni LV, Ursi M, Marasco G, Roberto M, Vestito A, Dajti E, Garcovich M, Bramanti S, Taurino D, Quagliarella F, Ciceri F, Prete A, Pession A, Festi D; ELASTOVOD Study Group; Bonifazi F. Diagnostic accuracy of liver stiffness measurement for the diagnosis of veno-occlusive disease/sinusoidal obstruction syndrome after hematopoietic stem cell transplantation (HSCT), the ELASTOVOD STUDY: an investigator-initiated, prospective, multicentre diagnostic clinical trial. Bone Marrow Transplant. 2025 Jul;60(7):978-993. doi: 10.1038/s41409-025-02570-w. Epub 2025 Apr 19. PMID 40253530